CLINICAL TRIAL: NCT06986577
Title: Evaluation of Mechanical Ventilation Methods Applied During the Procedure in Pediatric Cardiac Radiofrequency Ablation Interventions: Prospective Observational Study
Brief Title: Effect of Mechanical Ventilation on Cardiac RF Ablation
Status: Active, not recruiting | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Gözde Gürsoy Çirkinoğlu, MD, Izmir City Hospital
Other Study IDs: Mechanical Ventilation
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-01

CONDITIONS: Radiofrequency Catheter Ablation
Keywords: mechanical ventilation; cardiac radiofrequency ablation; pediatric arryhtmia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1) Lung protective mechanical ventilation: Mechanical ventilation with 7-9 ml tidal volume during RF
- 2) Low tidal volume high frequency ventilation: Mechanical ventilation with 4 ml tidal volume with high frequency during RF
- 3) Apnea ventilation: Apne ventilastion during RF

SUMMARY:
The aim of this study is to describe the results of cardiac radiofrequency ablation under general anesthesia.

to evaluate mechanical ventilation methods in pediatric patients. The main questions it aims to answer are

1. Whether lower tidal volume high frequency mechanical ventilation effects the success of radiofrequency ablation in pediatric cardiac arryhtmia patient?
2. The effect of mechanical ventilation strategies on the number of effective lesions, radiofrequency ablation time and arrhythmia recurrence in the first month

DETAILED DESCRIPTION:
Radiofrequency ablation (RF) is an effective method for the threatment of cardiac arrhythmias in pediatric patients. General anaesthesia and mechanical ventilation is the most common anesthesia management for pediatric arrhythmia patients. During the prosedure, thoracic excursion results in displacement of the catheter and disrupts the catheter stability which is crucial for quality of contact force (CF), sufficient ablation and safety. To minimize the thoracic excursion, high frequency low tidal volume ventilation and apnea ventilation may be needed during radiofrequency ablation. According to investigators knowledge there are studies about ventilatory strategies in adult patients who underwent cardiac radiofrequency ablation. However, there are no studies corcerning pediatric patients. In this study investigators aimed to investigate best ventilatory strategy for minimize thoracic excursion in pediatric patients with general anaesthesia. In this study investigators are going to observe 3 different ventilation strategies on radiofrequency ablation.

1. Lung protective mechanical ventilation with 7-9 ml/kg tidal volume,
2. Low tidal volume (4 ml/kg) high frequency mechanical ventilation
3. Apnea ventilation during radiofrequency ablation

ELIGIBILITY:
Inclusion Criteria:

* Between 0-18 years
* Paediatric surgery under general anaesthesia at Izmir City Hospital in the last 3 months since the date undergoing cardiac radiofrequency ablation procedure
* Procedures were performed with catheters with contract force measurement feature patients with

Exclusion Criteria:

* Patients with maintenance other than inhalation anaesthesia
* Patients whose anaesthesia method is changed during the procedure
* Patients with airway complications
* Development of haemodynamic instability during the procedure
* Patient with a history of previous cardiac surgery
* Presence of additional cardiac disease, advanced connective tissue disease, connective tissue disease, mitochondrial muscle disease

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: During the 3-month period, cardiac paediatric patients undergoing radiofrequency ablation under general anaesthesia in the catheterisation laboratory will be analysed
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Contact force | intraprosedural
  continuously measured through the catheter

SECONDARY OUTCOMES:
Lession count | intraprosedural
  number of successful lesions
Time | intraprosedural
  RF time

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Gürsoy Çirkinoğlu, MD, Principal Investigator — Izmir City Hospital, Anesthesiology and Reanimation Department; Halide Hande Sahinkaya, MD, Study Chair — Izmir City Hospital, Anesthesiology and Reanimation Department; Zeki Tuncel Tekgül, Prof. Dr., Study Chair — University of Health Sciences, Izmir City Hospital, Anesthesiology and Reanimation Department; Cem Karadeniz, Prof. Dr, Study Chair — Izmir Katip Celebi University Medical Faculty, Pediatric Cardiology Department
Locations (1):
- İzmir City Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Osorio J, Varley A, Kreidieh O, Godfrey B, Schrappe G, Rajendra A, Silverstein J, Romero J, Rodriguez D, Morales G, Zei P. High-Frequency, Low-Tidal-Volume Mechanical Ventilation Safely Improves Catheter Stability and Procedural Efficiency During Radiofrequency Ablation of Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2022 Apr;15(4):e010722. doi: 10.1161/CIRCEP.121.010722. Epub 2022 Mar 25. No abstract available. PMID 35333095
- [Result] Sivasambu B, Hakim JB, Barodka V, Chrispin J, Berger RD, Ashikaga H, Ciuffo L, Tao S, Calkins H, Marine JE, Trayanova N, Spragg DD. Initiation of a High-Frequency Jet Ventilation Strategy for Catheter Ablation for Atrial Fibrillation: Safety and Outcomes Data. JACC Clin Electrophysiol. 2018 Dec;4(12):1519-1525. doi: 10.1016/j.jacep.2018.08.016. Epub 2018 Nov 1. PMID 30573114
- [Result] Janson CM, Shah MJ, Kennedy KF, Iyer VR, Sweeten TL, Glatz AC, Steven JM, O'Byrne ML. Comparison of Outcomes of Pediatric Catheter Ablation by Anesthesia Strategy: A Report From the NCDR IMPACT Registry. Circ Arrhythm Electrophysiol. 2021 Jul;14(7):e009849. doi: 10.1161/CIRCEP.121.009849. Epub 2021 Jun 17. PMID 34137629